CLINICAL TRIAL: NCT03774238
Title: Biological and Functional Determinants of the Endothelial and Vascular Response to Exercise Training in COPD Patients
Brief Title: Determinants of the Vascular Response to Training in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: cDysEndoBPCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analyses will be carried out with the recruited population.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL18_0439; 2018-A02886-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-10-30; First posted 2018-12-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-02

CONDITIONS: COPD Patients; Healthy
Keywords: Flow-mediated dilatation; COPD; Pulmonary Rehabilitation; Comorbidities; endothelial cell; oxidative stress
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Masking Description: COPD patient group (n=50) and Healthy control Group (n=24)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD patients (Experimental): FMD analysis Endothelial progenitors Exercise test Exercise training
  Interventions: Other: FMD analysis
- Healthy subject (Experimental): FMD analysis Endothelial progenitors Exercise test
  Interventions: Other: FMD analysis

INTERVENTIONS:
Other: FMD analysis — Blood sample and vascular exploration.

SUMMARY:
Vascular comorbidities constitute a major burden in COPD patients. The atherosclerosis process is preceded by the onset of an endothelial dysfunction (assessed by the flow-mediated dilatation (FMD)), which is a risk factor for later ischemic vascular complications and death. In COPD, this endothelial dysfunction could be explained by intrinsic endothelial cell properties, or the effect of a pathogenic endothelial cell microenvironment (inflammation and/or oxidative stress). Exercise training constitue a powerful stimulus for the endothelial function, and could be mediated by the mobiliaztion and function of endothelial progenitors. While exercise training is an efficient intervention in COPD patients, its vascular effect appear blunted. The endothelial function response to training has appeared heterogeneous in COPD patients, and possibly linked to the endothelial cel lesion. Thus, endothelial function (assessed by the FMD) response to exercise training would be lower in COPD patients with a baseline impairment of the their FMD. In addition, of biological and functional factors could explained the magnitude of the FMD response in COPD patients.The aim of the study are thus :

To compare the FMD change in COPD patients with FMD above (FMD+) and under the median FMD (FMD-) after 4 weeks of exercise training in the whole study population.

To compare between COPD patients FMD+, COPD patients FMD- and healthy "control" subjects, the endothelial inflammation and senescence at baseline and the endothelial progenitor mobilization and function change induced by exercise (maximal exercise test and training).

To compare between COPD patients FMD+, COPD patients FMD- and healthy "control" subjects the effect of the endothelial microenvironment on the cellular pathways regulating the endothelial function in vitro at baseline and changes after exercise training.

To test in COPD patients the association between the magnitude of the FMD changes after training and biological, functional and clinical factors (inflammation oxidative stress markers, endothelial biomarkers, pulmonary impairment and phenotype, cardiovascular risks factors, vascular function, metabolic markers, physical activity level, …)

ELIGIBILITY:
Inclusion Criteria:

A/ COPD patients

* age between 35 and 85 years old
* spirometry showing an FEV1/VC < lower limit of normal
* with an indication for a pulmonary rehabilitation program
* written and informed consent for this study signed by the patient

B/ Healthy subjects

* age between 35 and 85 years old
* no cardiovascular or respiratory disease
* normal spirometry

Exclusion Criteria:

* Unstabilized comorbidity
* Subject in a period of exclusion relative to another protocol
* Major protected by law
* Subject participating in another research protocol
* Subject not affiliated to a social security scheme
* Pregnant or lactating woman
* Patient deprived of freedom by court or administrative order

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Measure of Flow-Mediated Dilatation (FMD) | post exercise and after 4 +/- 2 weeks of training
  Measure of FMD by EndoPAT2000©

SECONDARY OUTCOMES:
Measure of biological vascular markers | after 4 +/- 2 weeks of training
  E-selectin soluble (sE-sel), endotheline 1 (ET1), facteur von Willebrand (vWF), vascular endothelial growth factor A (VEGF-A), Fms-like tyrosine kinase receptor 1 soluble (sFlt-1), Angiopoietine 1 et 2 (Ang-1 Ang-2)
Number of colonies and function of Endothelial-Colony Formaing cells (ECFC) in vitro | post exercise and after 4 +/- 2 weeks of training
Number endothelial progenitors | post exercise and after 4 +/- 2 weeks of training
  CD34+, CD45+ and KDR + subpopulations by flow cytometry
Vascular function parameters | after 4 +/- 2 weeks of training
  Systolic pressure index (in AU)
Vascular function parameters | after 4 +/- 2 weeks of training
  Intima-media thickness (in mm)
Vascular function parameters | after 4 +/- 2 weeks of training
  Pulse-wave velocity (in ms-1)
Pulse-wave velocity (in ms-1) | after 4 +/- 2 weeks of training
Markers of systemic inflammation | after 4 +/- 2 weeks of training
  C-Reactive protein (in ng/ml)
Markers of oxidative stress | after 4 +/- 2 weeks of training
  Lipid peroxidation (in micromol/L)
Muscle function parameters | after 4 +/- 2 weeks of training
  Maximum isometric voluntary contraction (in N.m)
Exercise capacity and vascular adaptation parameters | after 4 +/- 2 weeks of training
  Maximal oxygen uptake (VO2max, in mL/kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Fares Gouzi, MD, PhD, Principal Investigator — UH Montpellier
Locations (2):
- France (2):
  - CHU Montpellier and CHU Nimes, Montpellier
  - University Hospital, Paris, Paris

IPD SHARING:
Plan to Share IPD: No